CLINICAL TRIAL: NCT00421746
Title: A Proof of Biological Efficacy Study Assessing the Potential of Piboserod, a Specific 5-HT4 Antagonist, for the Treatment of Symptomatic Congestive Heart Failure on Top of Usual Evidence Based Pharmacological Treatment
Brief Title: A Clinical Study Assessing the Potential of Piboserod for the Treatment of Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bio-Medisinsk Innovasjon (Industry)
Collaborators: Smerud Medical Research International AS (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMI 001 / SMR-1389
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — piboserod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Piboserod

SUMMARY:
The purpose of this study is to determine whether piboserod, a serotonin-4 receptor antagonist, is effective for the treatment of patients with congestive heart failure.

DETAILED DESCRIPTION:
Despite intensive research for decades, mortality and morbidity in chronic heart failure remains quite high. There is an obvious need for new drugs, especially drugs which may have a different mode of action than the existing ones on the market.

The purpose of this trial is to evaluate whether a new drug candidate, piboserod, has beneficial biological effects in stable outpatients with symptomatic heart failure receiving evidence based treatment for heart failure and to assess safety and tolerability of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CHF (NYHA class II-IV)
* Locally determined LVEF < 0.35 (by CMR, echocardiography, LV angiography, or radionuclide cardioangiography)
* Stable sinus rhythm
* Stable evidence based pharmacological treatment for CHF.

Exclusion Criteria:

* Unstable patients hospitalised within last 2 weeks
* Baseline prolongation of QTc interval
* Atrial fibrillation at randomisation
* MI or re-vascularisation last 3 months
* Stroke last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2006-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end-of-therapy in Left Ventricular Ejection Fraction, as measured using CMR imaging | 6 months

SECONDARY OUTCOMES:
Change in LV systolic and diastolic volume (and/or diameter) by CMR | 6 months
Change in NYHA functional class | 6 months
Change in various biomarkers for heart failure | 6 months
Change in QoL-scores | 6 months
Change in 6-minute walk distance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Torp-Pedersen, Dr. Med, Study Chair — Bispebjerg Hospital
Locations (17):
- Denmark (8):
  - Rigshospitalet, Copenhagen
  - Amager Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Amtsygehuset i Herlev, Herlev
  - Hvidovre Hospital, Hvidovre
  - Odense Universitets Hospital, Odense
  - Svendborg Sygehus, Svendborg
- Norway (6):
  - Østlandske Hjertesenter, Moss
  - Fana Hjertesenter, Nesttun
  - Rikshospitalet, Oslo
  - Ullevål Universitetssykehus, Oslo
  - Stavanger Universitetssjukehus, Stavanger
  - St. Olavs Hospital, Trondheim
- United Kingdom (3):
  - Castel Hill Hospital, Cottingham, East Yorkshire
  - Bridlington and District General Hospital, Bridlington
  - Western Infirmary, Glasgow

REFERENCES:
- [Derived] Kjekshus JK, Torp-Pedersen C, Gullestad L, Kober L, Edvardsen T, Olsen IC, Sjaastad I, Qvigstad E, Skomedal T, Osnes JB, Levy FO. Effect of piboserod, a 5-HT4 serotonin receptor antagonist, on left ventricular function in patients with symptomatic heart failure. Eur J Heart Fail. 2009 Aug;11(8):771-8. doi: 10.1093/eurjhf/hfp087. Epub 2009 Jun 30. PMID 19567409
- See also: Sponsor's web site — http://www.bmioslo.no